CLINICAL TRIAL: NCT03632980
Title: Evaluation of a Dynamic Focusing Ultrasonic Transducer for High Intensity Focused Ultrasound (HIFU) Treatment of Localized Prostate Adenocarcinoma - Dose Escalation Trial to Define the Best Acoustic Parameters
Brief Title: Dynamic Focusing Evaluation for Prostate Cancer Treatment
Acronym: FOC/DYN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: EDAP TMS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/F/10.08; 2011-A00313-38 (Other: AFSSAPS)
Record Dates: First submitted 2012-01-31; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Cancer of Prostate
Keywords: HIFU; Localized Prostate cancer; MRI; PSA nadir; Biopsy; High Intensity Focused Ultrasound; Prostate Specific Antigen (PSA)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIFU prostate treatment (Experimental): The HIFU intervention will concern Primary care patients or Secondary care patients (salvage).
  Intervention with "Ablatherm Foc/Dyn" or "Focal One" HIFU treatment devices
  HIFU intervention will be administered with "Ablatherm Foc/Dyn or Focal One - First line" to Patients suffering from localized prostate cancer that has not been previously treated or Salvage HIFU intervention will be administered with "Ablatherm Foc/Dyn or Focal One - Post radiotherapy" to subjects harboring prostate cancer recurrency after radiotherapy
  Interventions: Device: "Ablatherm Foc/Dyn" or "Focal One" HIFU treatment

INTERVENTIONS:
Device: "Ablatherm Foc/Dyn" or "Focal One" HIFU treatment — Non invasive treatment of localized prostate cancer by High Intensity Focused Ultrasound therapy, endorectal application.
  or Non invasive treatment of localized prostate cancer recurrency by High Intensity Focused Ultrasound therapy after radiotherapy failure, endorectal application.
  Other Names: Ablatherm Foc/Dyn or Ablatherm Foc/Dyn post-radiotherapy; Focal One or Focal One post-radiotherapy; First line treatment or Salvage treatment post-radiotherapy

SUMMARY:
Define the best acoustic parameters for the dynamic focusing HIFU transducer in the treatment of localized Prostate Cancer.

ELIGIBILITY:
Inclusion Criteria for primary care patients:

* Age > 70 years
* T1 or T2
* PSA < 15 ng/mL
* 12 randomized biopsies
* Gleason score ≤ 3+4
* Normal anal and rectal anatomy
* American Society of Anesthesiologists risk (ASA) 1 or 2

Exclusion Criteria for primary care patients:

* T3 patients
* American Society of Anesthesiologists risk (ASA) 3
* Metastatic disease (Bone scan…)
* Previous prostate cancer therapy
* Distance between rectal mucosa and prostatic capsule of more than 8 mm thickness
* Prostate volume over 50cc
* Previous bladder cancer
* contraindication to MRI
* previous rectal or urinary fistulae

Inclusion Criteria for salvage patients:

* Age > 50 years
* T1 or T2
* Biochemical recurrence after radiotherapy (Phoenix definition: nadir+2ng/ml)
* 12 randomized biopsies
* Normal anal and rectal anatomy
* ASA 1 or 2

Exclusion Criteria for salvage patients:

* T3 patients
* ASA 3
* Metastatic disease (Bone scan…)
* Distance between rectal mucosa and prostatic capsule of more than 8 mm thickness
* Prostate volume over 50cc
* Previous bladder cancer
* contraindication to MRI
* previous rectal or urinary fistulae

Min Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-06; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Necrosis measurement (immediate efficacy) | Day 7
  The coagulation necrosis induced by the HIFU dynamic focusing treatment of the prostate is evaluated by MRI in the first week post treatment.

SECONDARY OUTCOMES:
Histological marker measurement (mid term efficacy) | 6 months
  The mid term efficacy is evaluated by the rate of negative biopsy at 6 months.
Biochemical marker measurement (mid term efficacy) | 6 months
  The mid term efficacy is evaluated by the percentage of patient with a PSA nadir ≤ 0.3ng/mL
Rectal wall preservation (immediate safety and morbidity) | Day 7
  Evaluate the rectal wall preservation by MRI in the first week post treatment.
Adverse events reporting rates (safety and the morbidity) at 6 months | 6 months
  Adverse Events reporting
Adverse events reporting rates (safety and the morbidity) at 24 months | 24 months
  Adverse Events reporting
Quality of life score | 3 months
  Quality of life will be assessed using the QLQC30 (Quality of Life questionnaire) questionnaire.
  It is a specific questionnaire to determine the quality of life a patient with cancer. It is composed of 30 questions with 4 potential answers going from: not at all, a little, enough or a lot, within 28 questions and with a visual scale going from 1 to 7 (7 being excellent and 1 being very bad) for the last 2 questions. The raw score is established by adding the score of each question and a linear transformation range it from 0 to 100. The higher the score, the worse the quality of life.
Quality of life score | 6 months
  Quality of life will be assessed using the QLQC30 (Quality of Life questionnaire) questionnaire.
  It is a specific questionnaire to determine the quality of life a patient with cancer. It is composed of 30 questions with 4 potential answers going from: not at all, a little, enough or a lot, within 28 questions and with a visual scale going from 1 to 7 (7 being excellent and 1 being very bad) for the last 2 questions. The raw score is established by adding the score of each question and a linear transformation range it from 0 to 100. The higher the score, the worse the quality of life.
IPSS score | 3 months
  Urinary function will be assessed using the IPSS (International Prostate Score Symptom) questionnaire.
  The IPSS questionnaire is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35. The score is then categorized as follow: Mild (symptoms score less than or equal to 7), Moderate (symptom score range 8-19), Severe (symptom score range 20-35). The higher the score, the worse the symptoms.
IPSS score | 6 months
  Urinary function will be assessed using the IPSS (International Prostate Score Symptom) questionnaire.
  The IPSS questionnaire is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35. The score is then categorized as follow: Mild (symptoms score less than or equal to 7), Moderate (symptom score range 8-19), Severe (symptom score range 20-35). The higher the score, the worse the symptoms.
IIEF-5 score | 3 months
  Sexual function will be assessed using the IIEF-5 (The International Index of Erectile Function) questionnaire.
  The IIEF-5 Questionnaire is composed of 5 items with 5 possible answers rating from 1 to 5 (very low, low, moderate, high, very high).
  The score is the sum of the ordinal responses to the 56 items. It is then categorized as follow: 22-25: No erectile dysfunction, 17-21: Mild erectile dysfunction, 12-16: Mild to moderate erectile dysfunction, 8-11: Moderate erectile dysfunction, 5-7: Severe erectile dysfunction. The higher the score, the better the sexual function.
IIEF-5 score | 6 months
  Sexual function will be assessed using the IIEF-5 (The International Index of Erectile Function) questionnaire.
  The IIEF-5 Questionnaire is composed of 5 items with 5 possible answers rating from 1 to 5 (very low, low, moderate, high, very high).
  The score is the sum of the ordinal responses to the 56 items. It is then categorized as follow: 22-25: No erectile dysfunction, 17-21: Mild erectile dysfunction, 12-16: Mild to moderate erectile dysfunction, 8-11: Moderate erectile dysfunction, 5-7: Severe erectile dysfunction. The higher the score, the better the sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Albert GELET, MD, Principal Investigator — Edouard Herriot Hospital, Lyon, France
Locations (1):
- Edouard Herriot Hospital, Lyon, France